CLINICAL TRIAL: NCT07177547
Title: Screening and Referral Practices for Anxiety and Depression Among Patients With Chronic Neck, Shoulder and Low Back Pain Within Private Physiotherapy Practices: a Qualitative Study.
Brief Title: Screening and Referral Practices for Anxiety and Depression Among Patients With Chronic Neck, Shoulder and Low Back Pain Within Physiotherapy Practices
Status: Active, not recruiting | Type: Observational
Sponsor: Ana Catarina Navarro Ramalho (Other)
Responsible Party: Sponsor-Investigator, Ana Catarina Navarro Ramalho, PhD researcher, Department of Rehabilitation Sciences, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: S69684
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Chronic Musculoskeletal Pain; Anxiety; Depression
Keywords: Physiotherapy; Chronic musculoskeletal pain; Anxiety; Depression; Screening; Referral; Qualitative study
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Physical Therapy Modalities; Mass Screening; Referral and Consultation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mental health screening and referral practices in physiotherapy — Semi-structured interviews were conducted with 18 physiotherapists working in private settings to explore recognition, screening, and referral practices for anxiety and depression in patients with chronic musculoskeletal pain.
  Other Names: Screening for anxiety and depression in private physiotherapy practice; Screening for anxiety and depression in private physiotherapy practice Physiotherapist-led mental health recognition and referral

SUMMARY:
The goal of this cross-sectional, qualitative study is to investigate whether physiotherapists screen for symptoms of anxiety and depression in patients with chronic musculoskeletal pain and to explore the facilitators and barriers related to these practices. The main questions aim to answer are:

* What are the current practices of physiotherapists in private practice for screening anxiety and depression among patients with chronic musculoskeletal pain?
* What are the facilitators and barriers influencing physiotherapists' screening and referral practices for mental health care?

Participants will:

* Take part in a semi-structured interview (online or in person).
* Be asked about their experiences, attitudes, and practices related to recognizing, screening, managing, and referring patients with anxiety and depression.
* Participants will share perspectives on barriers and facilitators to integrating mental health screening into physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

- Physiotherapists treating patients with chronic musculoskeletal conditions.

Purposive sampling was used to obtain:

* Varied clinical experience: Less than 5 years of practice and more than 5 years of practice.
* Varied exposure to mental health training: With and without specialized training in mental health.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physiotherapists working in private practice settings in Belgium, with variation in gender, years of clinical experience, and prior mental health training.
  Recruitment was conducted through two channels:
  * Open-access contact list on the website of Axxon, the official Belgian physiotherapy professional association;
  * Direct outreach to physiotherapists who had previously completed mental health-related training and consented to future research contact.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Physiotherapists' perspectives on screening and referral practices for anxiety and depression symptoms in patients with chronic musculoskeletal pain. | From study start until completion of interviews and data analysis (approximately 6 months)
  Themes identified through qualitative framework analysis of semi-structured interviews with 18 physiotherapists. The analysis focuses on recognition, screening, management, and referral practices for anxiety and depression in patients with chronic musculoskeletal pain, including barriers, facilitators, and professional experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- Axxon website, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No